CLINICAL TRIAL: NCT01559246
Title: Comparison of Short Term Holter Monitoring vs. Long Term Zio(R)Patch True Continuous ECG Monitoring (TCEM Study)
Brief Title: True Continuous ECG Monitoring (TCEM Study)
Acronym: TCEM
Status: Completed | Type: Observational
Sponsor: iRhythm Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: iRT-001-2012
Record Dates: First submitted 2012-03-09; First posted 2012-03-21 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cardiac Arrhythmia
Keywords: Cardiac Arrhythmia Monitoring; Holter Monitoring; Continuous ECG monitoring; Event monitoring; Observational
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Arrhythmia: Subjects 18 years of age or greater that have indications for traditional cardiac(Holter) monitoring.

SUMMARY:
The purpose of this study is to compare short term (up to 48 hours) traditional cardiac rhythm monitoring using a standard ambulatory Holter monitor versus long term (up to 14 days), continuous ambulatory cardiac rhythm monitoring using a new device cleared by the FDA (Zio® Patch), iRhythm Technologies, Inc., San Francisco CA) in patients with suspected cardiac arrhythmias.

DETAILED DESCRIPTION:
This is a prospective, observational study of patients seen in the Holter lab at Scripps Green Hospital and other Scripps Clinic locations. Only patients who have indications for traditional cardiac rhythm monitoring will be enrolled in the study. Patients 18 years or older with suspected arrhythmias capable of providing informed consent will wear both a traditional Holter monitor for up to 48 hours and a Zio® Patch for up to 14 days. Both devices will be initiated at the same time as they do not interfere with one another. This will also allow a direct comparison of the same initial up to 24 hour monitoring period between the two devices. As the Zio® Patch is worn for up to 14 days instead of only 24 hours, it will be assessed if in the physician's opinion (referring physician), waiting for the extended time hinders being able to provide medical care and/or diagnosis for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Are being seen in the outpatient office for evaluation, treatment, or follow-up of arrhythmias;
* Have a medical history for which ascertaining whether asymptomatic arrhythmias is occurring could be helpful in their treatment plan;
* Are capable of giving informed consent; assessed by the investigator or the Study Coordinator;
* Are 18 years of age or older;
* Able to comply with long term continuous monitoring ECG device.

Exclusion Criteria:

* Have known skin allergies, conditions, or sensitivities (e.g. allergy to adhesives, psoriasis) as the Zio(R)Patch should not be used on patients with known skin allergies, conditions, or sensitivities; or
* Are receiving pacing therapy (e.g., from a pacemaker); or
* Are anticipated to receive or require external cardiac defibrillation during the monitoring period; or
* Are anticipated to be exposed to high frequency surgical equipment during the monitoring period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age of greater with suspected arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Arrhythmia detection for Zio® patch and the traditional ambulatory Holter monitor. | Up to 14 days.
  Data will be examined to determine the difference in the number of 6 types of arrhythmias detected at maximum observation times of 14 days and 24 hours respectively. In comparing the difference of the number of arrhythmias for the Zio® Patch and the Holter data, we are expecting a skewed distribution of the differences and will use a paired Wilcoxon Signed Rank Test since the normality assumption is not met for a paired t-test. If the difference is significantly greater than zero, there is evidence that the Zio® Patch is an improvement in this sample.

SECONDARY OUTCOMES:
Subjects ease in comfort for the Zio® Patch and the traditional ambulatory Holter monitor. | Up to14 days.
  Subjects will be given surveys to complete at different time points. Surveys to include questions assessing subjects preference in devices. McNemar's Test will be used to examine if the responses for ease of wear was different between the Zio® Patch and the Holter. Comparing both devices when the Holter is returned in the first 24/48 hours, and comparing the Holter at 24/48 hours and the Zio® Patch at total observation (up to 14 days). McNemar's Test will be used to compare if the patient would use the Zio® Patch again and if they would use the Holter.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Health, La Jolla, California, United States

REFERENCES:
- [Derived] Barrett PM, Komatireddy R, Haaser S, Topol S, Sheard J, Encinas J, Fought AJ, Topol EJ. Comparison of 24-hour Holter monitoring with 14-day novel adhesive patch electrocardiographic monitoring. Am J Med. 2014 Jan;127(1):95.e11-7. doi: 10.1016/j.amjmed.2013.10.003. Epub 2013 Oct 15. PMID 24384108